CLINICAL TRIAL: NCT03874312
Title: Ultrasound-assessed Internal Jugular Vein Distensibility to Predict Right Atrial Pressure and Other Hemodynamic Parameters in Patients With Advanced Chronic Heart Failure
Brief Title: Ultrasound-assessed Internal Jugular Vein Distensibility in Advanced Chronic Heart Failure (US-IJVD in CHF)
Acronym: US-IJVD-CHF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 371-072017
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Systolic Chronic Heart Failure; Congestion, Venous; Advanced Heart Failure
Keywords: right heart catheterization; Peripheral congestion; Right atrial pressure; Internal jugular vein distention ratio; ultrasound of jugular vein; chronic heart failure
MeSH Terms: conditions — Hyperemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Calibration group: Patients with systolic chronic heart failure who undergo right heart catheterization (RHC) for heart transplant/left ventricular assist device workup.
  Interventions: Diagnostic Test: Linear ultrasound (US) assessment of the internal jugular vein
- Validation group: Patients with systolic chronic heart failure who undergo RHC for heart transplant/left ventricular assist device workup.
  Interventions: Diagnostic Test: Linear ultrasound (US) assessment of the internal jugular vein

INTERVENTIONS:
Diagnostic Test: Linear ultrasound (US) assessment of the internal jugular vein — Evaluation of jugular vein distensibility at rest and after Valsalva maneuver by US at the time of the RHC. US-guided IJV is routinely performed at the time of vein cannulation.

SUMMARY:
Prospective validation of the ultrasound-assessed internal jugular vein distensibility (JVD) ratio to identify patients with systolic chronic heart failure and right atrial pressure (RAP) of 7 or less mmHg measured by the right heart catheterization. In a calibration cohort, a threshold ratio will be identified, above which the RAP is normal with the highest accuracy. This diagnostic tool with a defined threshold of the JVD ratio will be assessed in a second prospective validation cohort.

DETAILED DESCRIPTION:
Peripheral congestion is caused by an excess of fluid in tissues and vessels. Fluid overload is associated with poor outcome in heart failure (HF)(1). Several clinical signs can suggest peripheral congestion, such as peripheral edema or neck vein distention. In particular, the clinical sign of the neck jugular vein distention is used to estimate right atrial pressure (RHC) and is associated with fluid overload and congestion. Nevertheless, clinical assessment is somewhat subjective depending on the anatomy of the patient's neck and on the expertise of the physician (2). It has been reported that the detection of elevated RAP can be measured using a bedside ultrasound (US)(3). In this study, the Authors compared the jugular vein distensibility (IVD) ratio assessed with US with the invasive measure of the RAP reporting a good accuracy in detecting normal RAP. They showed a good performance of this diagnostic test, nevertheless, they evaluated this diagnostic test in a mix population including only 27 patients with congestive HF. More recent studies showed the prognostic value of the IVD ratio in patients with HF (4). Nevertheless, a specific threshold of the internal JVD ratio to identify patients with normal RAP in the setting of patients with systolic chronic HF (CHF) has never been described. Furthermore, in patients with CHF clinical signs of congestion cannot always be evident at clinical examination, making the decision to modify diuretic dosage or to introduce vasodilator drugs uneasy. Thus, a convenient, accurate, and reproducible non-invasive tool to identify patients with normal RAP (normal mean RAP is 7 or less mmHg) patients with systolic CHF would be desirable to tailor therapy, in particular in outpatient clinics.

The main hypothesis of this study is that US-assessment of the internal JVD could be an accurate diagnostic tool to identify patients with normal RAP in this challenging set of patients.

The primary aim of the study prospectively validates an US-assessed internal JVD ratio to identify patients with systolic CHF and RAP of 7 or less mmHg measured by RHC. In a calibration cohort, a threshold of the JVD ratio above which the RAP is normal with the highest accuracy will be identified and then this diagnostic tool with a defined JVD ratio will be validated in a second prospective validation cohort.

ELIGIBILITY:
Inclusion Criteria:

* All patients with systolic chronic heart failure defined by a left ventricular ejection fraction (LVEF) <50% on echocardiogram that, undergo elective RHC in the heart transplant/left ventricular assist device work-up.
* In case of occlusion of the left internal jugular vein (IJV), the RHC is performed from to contralateral IJV, and US-assessed JVD ratio will be measured on the right IJV.

Exclusion Criteria:

* Patients supported by a left ventricular assist device.
* Patients with acute heart failure that undergo RHC as an urgent procedure in hemodynamically unstable patients.
* Patients unable/unwilling to sign a written informed consent.
* Patients in which an RHC is not feasible from an internal jugular vein.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with systolic chronic heart failure defined by a left ventricular ejection fraction (LVEF) <50% on echocardiogram that, undergo elective RHC in the heart transplant/left ventricular assist device work-up.
  All procedure, RHC, ultrasound assessment of the IJV, echocardiogram, laboratory test exams are routine exams in the heart transplant/left ventricular assist device work-up or in the staging of patients with advanced HF. No adjunctive procedures have been performed for this specific study.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-10-18 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of patients with normal RAP (=<7 mmHg) with US-IJVD based on the JVD ratio obtained from the calibration cohort. | From July 2017 to June 2019
  Positive predictive value (PPV) of the JVD ratio to identify patients with normal (RAP=<7 mmHg) measured by RHC in the validation group. In particular a higher JVD ratio indicated lower RAP.

SECONDARY OUTCOMES:
Clinical major cardiac events among patients included in the calibration group divided on the basis of the JVD ratio | From July 2017 to June 2019
  Clinical events include cardiac death, unknown death, cardiac hospitalization, urgent heart transplant, left ventricular assist device implantation. In particular it is expected that patients with JVD ratio above the identified threshold in the calibration group have a better outcome.

OTHER OUTCOMES:
Relationship between JVD ratio and other hemodynamic parameters obtained by RHC | From July 2017 to June 2019
  The hemodynamic parameters will include pulmonary artery pressures and pulmonary capillary wedge pressure

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Ammirati, MD, PhD, Principal Investigator — Niguarda Hospital, Milano, Italy; Fabrizio Oliva, MD, Study Director — Niguarda Hospital, Milano, Italy; Davide Marchetti, MD, Study Chair — Università Statale di Milano, Italy; Andrea Garascia, MD, Study Chair — Niguarda Hospital, Milano, italy; Giada Colombo, Study Chair — Università Statale di Milano, Italy
Locations (1):
- De Gasperis Cardio Center, Niguarda Hospital, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
The informed consent does not include to make public the individual participant data

REFERENCES:
- [Background] Caldentey G, Khairy P, Roy D, Leduc H, Talajic M, Racine N, White M, O'Meara E, Guertin MC, Rouleau JL, Ducharme A. Prognostic value of the physical examination in patients with heart failure and atrial fibrillation: insights from the AF-CHF trial (atrial fibrillation and chronic heart failure). JACC Heart Fail. 2014 Feb;2(1):15-23. doi: 10.1016/j.jchf.2013.10.004. Epub 2014 Jan 8. PMID 24622114
- [Background] McGee SR. Physical examination of venous pressure: a critical review. Am Heart J. 1998 Jul;136(1):10-8. doi: 10.1016/s0002-8703(98)70175-9. PMID 9665212
- [Background] Simon MA, Kliner DE, Girod JP, Moguillansky D, Villanueva FS, Pacella JJ. Detection of elevated right atrial pressure using a simple bedside ultrasound measure. Am Heart J. 2010 Mar;159(3):421-7. doi: 10.1016/j.ahj.2010.01.004. PMID 20211304
- [Background] Pellicori P, Kallvikbacka-Bennett A, Dierckx R, Zhang J, Putzu P, Cuthbert J, Boyalla V, Shoaib A, Clark AL, Cleland JG. Prognostic significance of ultrasound-assessed jugular vein distensibility in heart failure. Heart. 2015 Jul;101(14):1149-58. doi: 10.1136/heartjnl-2015-307558. Epub 2015 May 25. PMID 26006717
- [Derived] Ammirati E, Marchetti D, Colombo G, Pellicori P, Gentile P, D'Angelo L, Masciocco G, Verde A, Macera F, Brunelli D, Occhi L, Musca F, Perna E, Bernasconi DP, Moreo A, Camici PG, Metra M, Oliva F, Garascia A. Estimation of Right Atrial Pressure by Ultrasound-Assessed Jugular Vein Distensibility in Patients With Heart Failure. Circ Heart Fail. 2024 Feb;17(2):e010973. doi: 10.1161/CIRCHEARTFAILURE.123.010973. Epub 2024 Feb 1. PMID 38299348